CLINICAL TRIAL: NCT00962936
Title: Phase I/II Study to Evaluate the Safety and Tolerability of the Monoclonal Antibody CT-011 in Patients With Chronic Hepatitis C Genotype I Infection
Brief Title: Safety and Tolerability Study of the Monoclonal Antibody CT-011 in Patients With Chronic Hepatitis C Genotype I Infection
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CureTech Ltd (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-2009-01
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; HCV Genotype I infection; Liver disease
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT-011 (Experimental)
  Interventions: Drug: CT-011

INTERVENTIONS:
Drug: CT-011 — CT-011

SUMMARY:
This study aims to evaluate whether an investigational monoclonal antibody, CT-011, is safe to give and if it helps patients with hepatitis C virus (HCV). Monoclonal antibodies are a type of drug that is typically given by infusion into a vein (intravenously). Results of this trial will help doctors obtain additional information with regard to the safety and efficacy of CT-011 as a potential treatment for HCV.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 60 years of age, both genders.
2. Biopsy proven infection with Hepatitis C genotype 1.
3. Positive for anti-HCV.
4. Chronically infected for at least 3 months from diagnosis.
5. ECOG performance status ≤ 1.
6. Previous therapy with interferon +/- Ribavirin or Peginterferon +/- Ribavirin or ineligibility for this type of therapy or for liver transplantation.

Exclusion Criteria:

1. Patients who received any type of anti viral treatment during the 3 months prior to enrollment.
2. Any history or active malignancy.
3. History of major organ transplantation with an existing functional graft.
4. Patients who received any systemic concurrent therapy within the last 4 weeks.
5. Patients progressing to acute liver failure (ALF).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of CT-011 in patients with Chronic Hepatitis C due to HCV Genotype I infection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel